CLINICAL TRIAL: NCT02896322
Title: Partial Breast Irradiation With Cyber Knife After Breast Conserving Surgery: A Pilot Study in Early Breast Cancer
Brief Title: Cyberknife After Breast Conservative Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INT 109/12
Record Dates: First submitted 2016-08-04; First posted 2016-09-12 (Estimated); Last update posted 2016-09-12 (Estimated); Status verified 2016-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

ARMS (1):
- Cyberknife (Experimental): APBI with cyberknife after breast conserving surgery in breast cancer
  Interventions: Radiation: Partial breast irradiation with cyberknife

INTERVENTIONS:
Radiation: Partial breast irradiation with cyberknife

SUMMARY:
Accelerated partial breast irradiation with CyberKnife (CK-APBI) is a promising innovative approach for early breast cancer after conservative surgery, for addressing the need of a radiotherapy target only to the surgical cavity in selected patients, exceeding the limits of other PBI/APBI.

DETAILED DESCRIPTION:
The large majority of local recurrences in breast cancer after breast conserving treatment are close to the original tumor site. This evidence suggested to restrict the radiotherapy target to the surgical cavity in selected patients. Consequently, shorter fractionation strategies focused only on tumor bed with a small cuff of surrounding subclinical disease, i.e. accelerated partial breast irradiation (APBI), were developed. Stereotactic radiotherapy was thought, consisting of a short course of intense treatment focused on the target tissue. There is very little experience with CiberKnife for early breast cancer until now.

This study is a prospective non-randomized study designed to assess the acute, sub-acute, late toxicity, cosmesis and globally the feasibility of CyberKnife (CK-APBI). From June 2013 to June 2018 we are going to enroll 80 patients considered eligible for the present study. All patients will be followed for at least 2 years. A first enrollment of 20-25 patients is scheduled as first assessment.

Breast magnetic resonance imaging (MRI) will be aided to mammography and ultrasound examination for confirming the best selection of patients.

For the assessment of acute toxicity, cosmetic results by three different observers (physician, patient, external observer), medium term and late toxicity, patients were evaluated and the results recorded immediately before and after radiotherapy, then after 1 month, three, six, nine, and twelve, and twenty-four months. The toxicity will be correlated to the main radiotherapy treatment dosimetry and delivery recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients were ≥45 years of age with stage I-IIA histologically confirmed breast carcinoma, with tumor-free (at least 2 mm or more) inked histologic margins at surgical resection.

Exclusion Criteria:

* Invasive lobular or multicentric carcinoma;
* Extensive associated non-invasive ductal carcinoma (synchronous or previous); peritumoral vascular invasion (>3 vessels);
* BRCA mutation carriers,
* >4 involved axillary lymph nodes,
* Distant metastasis,
* Non-epithelial malignancies of the breast,
* Synchronous contralateral invasive carcinoma,
* Paget disease,
* History of previous malignancy (except non-melanoma skin cancers and in situ oral cavity and cervix carcinoma);
* Further exclusion criteria were pregnancy, collagen vascular disease, aesthetic additive prostheses, severe cardiac, pulmonary and liver diseases, infectious, psychiatric illness compromising the correct acquisition of informed consent.

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2013-06; Primary Completion 2016-09 (Actual); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
acute and sub-acute toxicity according to NCI CTCAE Version 3.0 | within 6 months after the end of irradiation
  According to NCI CTCAE Version 3.0

SECONDARY OUTCOMES:
Late toxicity according to NCI CTCAE Version 3.0 | 24 months after the end of irradiation
  According to NCI CTCAE Version 3.0
Cosmesis according to NCI CTCAE Version 3.0 | 24 months after the end of irradiation
  According to NCI CTCAE Version 3.0

CONTACTS AND LOCATIONS:
Overall Officials: Laura Lozza, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Locations (2):
- Italy (2):
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Lombardy
  - Fondazione IRCCS Istituto Neurologico C. Besta, Milan, Lombardy

REFERENCES:
- [Derived] Lozza L, Fariselli L, Sandri M, Rampa M, Pinzi V, De Santis MC, Franceschini M, Trecate G, Maugeri I, Fumagalli L, Bonfantini F, Bianchi G, Pignoli E, De Martin E, Agresti R. Partial breast irradiation with CyberKnife after breast conserving surgery: a pilot study in early breast cancer. Radiat Oncol. 2018 Mar 23;13(1):49. doi: 10.1186/s13014-018-0991-4. PMID 29566762